CLINICAL TRIAL: NCT01836822
Title: Diagnostic Accuracy of Different Bronchoscopic Sampling Techniques in Patients With Mediastinal Lymph Node Enlargement Suspected of Sarcoidosis
Brief Title: Bronchoscopic Sampling Techniques in Sarcoidosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Rafał Krenke, MD, PhD, Medical University of Warsaw
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: IPU-DIMPA-WUM13(1)
Record Dates: First submitted 2013-04-17; First posted 2013-04-22 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Mediastinal Lymph Node Enlargement; Sarcoidosis; Tuberculosis; Lymphomas
Keywords: mediastinal lymph node enlargement; sarcoidosis; bronchoscopy; EBUS guided transbronchial needle aspiration (EBUS-TBNA); transbronchial needle aspiration (EBUS-TBNA); EBUS guided transbronchial forceps biopsy EBUS-TBFB)
MeSH Terms: conditions — Sarcoidosis; Tuberculosis; Lymphoma | interventions — Bronchoalveolar Lavage

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bronchoscopic lymph node sampling (Experimental): Several different sampling techniques will be used in each patient. They include: EBUS guided transbronchial needle aspiration (EBUS-TBNA), EBUS guided transbronchial forceps biopsy (EBUS-TBFB), large bore (19G) histologic needle biopsy of the mediastinal lymph nodes, forceps biopsy of bronchial mucosa in central and peripheral bronchi
  Interventions: Procedure: EBUS guided transbronchial forceps biopsy (EBUS-TBFB); Procedure: EBUS guided transbronchial needle aspiration (EBUS-TBNA); Procedure: large bore (19G) histologic needle biopsy of the mediastinal lymph nodes; Procedure: Bronchoalveolar lavage (BAL); Procedure: Endobronchial forceps biopsy

INTERVENTIONS:
Procedure: EBUS guided transbronchial forceps biopsy (EBUS-TBFB)
  Other Names: EBUS guided miniforceps biopsy
Procedure: EBUS guided transbronchial needle aspiration (EBUS-TBNA)
Procedure: large bore (19G) histologic needle biopsy of the mediastinal lymph nodes
Procedure: Bronchoalveolar lavage (BAL)
Procedure: Endobronchial forceps biopsy

SUMMARY:
The development of endobronchial ultrasound (EBUS) and EBUS-guided transbronchial needle aspiration (EBUS-TBNA) has improved the safety and diagnostic accuracy of the mediastinal lymph node (MLN) sampling. Still, in some diseases routine cytological specimens are considered insufficient and histological sampling is preferred. The aim of the study is to compare the diagnostic accuracy of EBUS-TBNA and two other, more invasive procedures to obtain histological samples from MLN in patients with clinical and radiological features of sarcoidosis.

Bronchoscopy with bronchoalveolar lavage (BAL), EBUS-TBNA, EBUS guided transbronchial forceps biopsy (EBUS-TBFB), large bore (19G) histology TBNA as well as endobronchial forceps biopsy will be performed in 90 consecutive patients with mediastinal lymph node enlargement and clinical and radiological features of sarcoidosis.

Diagnostic accuracy of each sampling technique will be calculated and compared to other techniques. Diagnostic yield of different technique combinations will also be calculated and the most efficient diagnostic approach will be defined.

ELIGIBILITY:
Inclusion Criteria:

* provided informed consent
* mediastinal lymph node enlargement that requires bronchoscopy and transbronchial sampling
* clinical presentation that might be consistent with sarcoidosis

Exclusion Criteria:

* age below 18 years
* known contraindications for bronchoscopy and/or mediastinal sampling, e.g. coagulation disorders
* lung or extrapulmonary tumors with suspicion of malignant mediastinal lymph node involvement

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-03 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Accuracy of different bronchoscopic sampling methods in making the diagnosis of sarcoidosis. | Approximately ten days after the procedure, when the results of the cytological and histopathological examination will be available
  Comparison of the diagnostic yield of the cytologic and histologic specimens collected by EBUS-TBNA, EBUS-TBFB, large bore TBNA, endobronchial forceps biopsy and BAL in terms of making the diagnosis of sarcoidosis.

SECONDARY OUTCOMES:
Adequacy of cytologic and histopathologic specimens collected by different sampling method as the diagnostic samples enabling confirmation of granulomatous lymph node disease. | up to 9 months
  Comparison of the number of patients in whom the specific sampling method has been undertaken (e.g. BAL, EBUS-TBNA, EBUS-TBFB and large bore TBNA) with the number of patients in whom the specific sampling method provided the adequate specimens, containing the elements of granulomas (also the relationship between the mediastinal lymph node dimension and the quality of the samples collected with different techniques)

OTHER OUTCOMES:
Local complications of mediastinal lymph node sampling | During and 24 hrs after bronchoscopic procedure
  The number of patients in whom mediastinal vessels would be injured (resulting in endobronchial or extrabronchial bleeding). The number of patients with pneumothorax and/or pneumomediastinum complicating mediastinal sampling

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Pneumonology and Allergology, Medical University of Warsaw, Warsaw, Poland